CLINICAL TRIAL: NCT01632761
Title: Effects of Vitamin D and Marine Omega-3 Fatty Acids on Anemia in the Elderly
Brief Title: Effects of Vitamin D and Marine Omega-3 Fatty Acids on Anemia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Office of Dietary Supplements (ODS) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Nancy Berliner, Chief, Hematology Division, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2012P001526
Record Dates: First submitted 2012-06-29; First posted 2012-07-03 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Anemia
Keywords: anemia; vitamin D3; omega-3 fatty acids; fish oil; primary prevention
MeSH Terms: conditions — Anemia | interventions — Cholecalciferol; Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin D + fish oil (Active Comparator): Dietary Supplement: Vitamin D3 (cholecalciferol), 2000 IU per day. Other Name: cholecalciferol Drug: omega-3 fatty acids (fish oil) Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Interventions: Dietary Supplement: Vitamin D3 .; Drug: omega-3 fatty acids (fish oil)
- Vitamin D + fish oil placebo (Active Comparator): Dietary Supplement: Vitamin D3 (cholecalciferol), 2000 IU per day. Other Name: cholecalciferol Dietary Supplement: Fish oil placebo Fish oil placebo
  Interventions: Dietary Supplement: Vitamin D3 .; Dietary Supplement: Vitamin D3 placebo
- Vitamin D placebo + fish oil (Active Comparator): Drug: omega-3 fatty acids (fish oil) Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Dietary Supplement: Vitamin D3 placebo Vitamin D placebo
  Interventions: Drug: omega-3 fatty acids (fish oil); Dietary Supplement: Fish oil placebo
- Vitamin D placebo + fish oil placebo (Active Comparator): Dietary Supplement:Vitamin D3 placebo Vitamin D placebo Dietary Supplement: Fish oil placebo Fish oil placebo
  Interventions: Dietary Supplement: Vitamin D3 placebo; Dietary Supplement: Fish oil placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 .
  Arms: Vitamin D + fish oil; Vitamin D + fish oil placebo
Drug: omega-3 fatty acids (fish oil)
  Arms: Vitamin D + fish oil; Vitamin D placebo + fish oil
Dietary Supplement: Vitamin D3 placebo
  Arms: Vitamin D + fish oil placebo; Vitamin D placebo + fish oil placebo
Dietary Supplement: Fish oil placebo
  Arms: Vitamin D placebo + fish oil; Vitamin D placebo + fish oil placebo

SUMMARY:
The VITamin D and OmegaA-3 TriaL (VITAL; NCT01169259) is a randomized clinical trial in 20,000 U.S. men and women studying whether taking daily dietary supplements of vitamin D3 (2000 IU) or omega-3 fatty acids (Omacor® fish oil, 1 gram) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. This ancillary study is being conducted among VITAL participants and will study whether vitamin D or fish oil: (A) in the overall VITAL cohort, reduces the number of persons diagnosed with anemia and (B) in a subcohort of 900 participants seen in Boston, effects long-term changes of the proteins in blood in both anemic and non-anemic individuals who provide blood samples at the start of the study and again 2 years later.

DETAILED DESCRIPTION:
The VITamin D and OmegA-3 Trial (VITAL; NCT01169259) is a randomized clinical trial of vitamin D (in the form of D3 [cholecalciferol]) and marine omega-3 fatty acid (eicosapentaenoic acid [EPA] + docosahexaenoic acid [DHA]) supplements in the primary prevention of cancer and cardiovascular disease.

Eligible participants will be assigned by chance (like a coin toss) to one of four groups: (1) daily vitamin D3 and omega-3; (2) daily vitamin D3 and omega-3 placebo; (3) daily vitamin D and omega-3; or (4) daily vitamin D placebo and omega-3 placebo. Participants have an equal chance of being assigned to any of these four groups and a 3 out of 4 chance of getting at least one active agent.

Participants in all group will take two pills each day--one softgel that contains either vitamin D3 or vitamin D placebo and one capsule that contains either omega-3 or omega-3 placebo. Participants will receive their study pills in convenient calendar packages via U.S. mail.

Participants will also fill out a short (15-20 minute) questionnaire each year. The questionnaire asks about health; lifestyle habits such as physical exercise, diet, and smoking; use of medications and dietary supplements; family history of illness, and new medical diagnoses. Occasionally participants may receive a phone call from study staff to collect information or to clarify responses on the questions.

If a participant reports a new medical diagnosis of anemia on the short questionnaires, he or she will be invited to participate in this sub-study. If the participant consents, his or her medical record will be reviewed to confirm the diagnosis of anemia. We expect roughly 1,100 individuals to develop anemia while on the study.

Of the expected 20,000 participants in the VITAL trial, approximately 1,000 participants will be seen in Boston and given the opportunity to participate in optional research blood draws. This sub-study expects to receive approximately 10mL of the samples collected from 900 of these participants. This portion of blood will be used to evaluate the amount of different proteins in both anemic and non-anemic individuals. Blood samples will be collected at baseline and two years later.

ELIGIBILITY:
Participants in VITAL (NCT 01169259) who do not have anemia at baseline and who report a diagnosis of anemia on the VITAL follow-up questionnaires are eligible to participate in this ancillary study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2012-11 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of Anemia | 2 years
  We will compare the number of participants who took vitamin D supplements who developed anemia and the number of participants who did not take vitamin D who developed anemia to current rates of development of anemia in the U.S. We will further examine whether the effect of vitamin D supplementation on anemia risk varies by race/ethnicity, gender, or baseline levels of 25(OH)D.
Long-term Changes in Blood Protein Levels | 2 years
  We will examine the samples from the 900 boston participants and determine whether vitamin D supplementation affects long-term changes in hemoglobin, red blood cell (RBC) indices, hepcidin, and erythropoietin (EPO) levels. These protein levels will be assessed in both anemic and non-anemic individuals in fresh samples at baseline [pre-randomization] and at 2 years of follow-up post-randomization.

SECONDARY OUTCOMES:
Incidence of Anemia | 2 years
  We will compare the number of participants taking fish oil supplements who developed anemia and the number of participants not taking fish oil supplements who developed anemia to the current rates of development of anemia in the U.S. We will also study the number participants diagnosed with anemia over 4 years of follow-up and whether the effect of taking fish oil supplements on anemia risk varies by race/ethnicity, gender, or baseline levels of omega-3 fatty acid.
Long-term Changes in Protein Levels | 2 years
  We will examine the samples collected from the 900 Boston participants and determine whether fish oil supplementation affects long-term changes in hemoglobin, red blood cell(RBC) indices, hepcidin, and erythropoietin (EPO) levels. These protein levels will be assessed in both anemic and non-anemic individuals in fresh samples at baseline [pre-randomization] and at 2 years of follow-up post-randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Berliner, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Welcome to the VITAL study website — http://www.vitalstudy.org/